CLINICAL TRIAL: NCT05543694
Title: ED90 of Epidural Bupivacaine for the Initiation of Labor Analgesia: A Randomized Biased Coin Sequential Allocation Trial With a Lidocaine Test Dose
Brief Title: ED90 of Epidural Bupivacaine With Lidocaine for the Initiation of Labor Analgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Associate Professor of Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022P002226
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Labor Pain; Analgesia
Keywords: Dural puncture epidural; Neuraxial Analgesia; Bupivacaine; Local Anesthetic
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial Using Biased Coin Design to Determine Effective Dose for 90% (ED90) of Subjects
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The biased-coin allocation after each successful response will be implemented by flipping a virtual biased coin (10% vs. 90% probability of randomizing the next patient to the lower vs. same dose than received by the last patient with the same epidural technique) using R statistical software (R Foundation for Statistical Computing, Vienna, Austria). Care Provider (Clinical Anesthesiologist) will administer the identified dose, then summon blinded observer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dural Puncture Epidural Technique (Experimental): Laboring women receiving the Dural Puncture Epidural (DPE) Technique, after a lidocaine "test dose", with dose of Bupivacaine 0.25% diluted to 20 mL with isotonic sterile 0.9% saline. The first subject in the DPE group will receive an initial dose of bupivacaine 25 mg, with an endpoint being the achievement of an NRS < 3 at 30 min. Subsequent patients are administered bupivacaine doses determined by the response of the previous subject, as per the biased coin method. The subsequent up and down interval doses are bupivacaine 2.5 mg (1 mL) increments, with an anticipated dose range from 20 mg to 40 mg.
  Interventions: Drug: Bupivacaine Hydrochloride
- Epidural Technique (Active Comparator): Laboring women receiving the Conventional Epidural Technique (EPL), after receiving a lidocaine "test dose" with dose of Bupivacaine 0.25% diluted to 20 mL with isotonic sterile 0.9% saline. The first subject in the EPL group will receive an initial dose of bupivacaine 25 mg, with an endpoint being the achievement of an NRS < 3 at 30 min. Subsequent patients are administered bupivacaine doses determined by the response of the previous subject, as per the biased coin method. The subsequent up and down interval doses are bupivacaine 2.5 mg (1 mL) increments, with an anticipated dose range from 20 mg to 40 mg.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Subjects will receive a dose of bupivacaine as described in the arm section of this trial

SUMMARY:
To estimate the dose of bupivacaine required to achieve initial effective comfort in 90% of patients (ED90) via the epidural (DPE or EPL) technique in women undergoing labor after receiving a lidocaine "test dose"

DETAILED DESCRIPTION:
The primary objective of our study is to use a biased coin up-down allocation methodology to estimate the dose of bupivacaine required to achieve initial effective comfort in 90% of patients (ED90) via the epidural (DPE or EPL) technique in women undergoing labor induction or augmentation; we hypothesize that we will be able to determine the ED90 of bupivacaine for each technique with adequate precision to inform the optimal doses. We will be conducting this study in women who receive a prior lidocaine "test dose" used in standard clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Parturient with no major co-morbidities
* Singleton, vertex gestation at term (37-42 weeks)
* Less than or equal to 5 cm dilation
* Desire to receive epidural labor analgesia
* Numerical Rating Scale greater or equal to 5 (NRS 0-10, where 0 = no pain, and 10 = worst pain imaginable), at time of epidural labor analgesia request.

Exclusion Criteria:

* Current or historical evidence of clinically significant disease or condition, including diseases of pregnancy (i.e preeclampsia, gestational diabetes)
* Any contraindication to the administration of an epidural technique
* History of hypersensitivity or idiosyncratic reaction to an amide local anesthetic agent
* Current or historical evidence of a disease which may result in the risk of a cesarean delivery (i.e. history of uterine rupture). NB: Exception-trial of labor after cesarean delivery (TOLAC) will be eligible.
* Evidence of anticipated fetal anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Verbal Numerical Pain Rating Score | 30 minutes
  (0-10, with higher scores meaning more pain); goal with analgesia is < 3/10

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngan Kee WD, Ng FF, Khaw KS, Lee A, Gin T. Determination and comparison of graded dose-response curves for epidural bupivacaine and ropivacaine for analgesia in laboring nulliparous women. Anesthesiology. 2010 Aug;113(2):445-53. doi: 10.1097/ALN.0b013e3181bdf9da. PMID 20613484
- [Background] Benhamou D, Ghosh C, Mercier FJ. A randomized sequential allocation study to determine the minimum effective analgesic concentration of levobupivacaine and ropivacaine in patients receiving epidural analgesia for labor. Anesthesiology. 2003 Dec;99(6):1383-6. doi: 10.1097/00000542-200312000-00022. PMID 14639153
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707